CLINICAL TRIAL: NCT06732063
Title: Evaluation of Postoperative Pain After Endodontic Retreatment Using Different Working Length Determination Methods: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: öznur dişli (Other)
Responsible Party: Sponsor-Investigator, öznur dişli, research assistant, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023/428
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: This Study Compares the Effects of Two Working Length Methods on Postoperative Pain in Single-rooted, Single-canal Teeth During Root Canal Retreatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Separate length determination method (Other)
  Interventions: Device: endodontic retreatment
- Simultaneous length determination method (Other)
  Interventions: Device: endodontic retreatment

INTERVENTIONS:
Device: endodontic retreatment — Re-treatment of previously failed root canal treatments

SUMMARY:
The aim of this study is to compare the effects of two different working length determination methods on the incidence of postoperative pain in single-rooted, single-canal teeth undergoing root canal retreatment (RCR). Sixty-four previously treated, single-rooted, single-canal teeth, which were determined to require RCR based on clinical symptoms and radiographic findings, were randomly and equally divided into two groups and included in the study. Two distinct working mechanisms of an integrated endodontic motor with an apex locator were used in our study. One method involved simultaneous determination of the working length during canal shaping, while the other method determined the working length with a hand file after the canal filling was removed. After the session in which the methods were applied and the working length was determined, participants' pain levels were recorded using a visual analog scale (VAS) at 6-12 hours and on days 1-2-3-4-5-6-7.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers aged between 18 and 65 with no systemic diseases. Teeth without acute apical abscess. Single-rooted and single-canal teeth that have previously undergone root canal treatment, failed, and require re-treatment (diagnosed based on clinical symptoms and radiographic findings).

Individuals with preoperative pain rated 50 or lower on the 100 mm VAS scale

Exclusion Criteria:

Individuals with systemic diseases or allergic reactions. Pregnancy and breastfeeding. Teeth with open apex. Teeth with internal or external root resorption. Patients who have taken analgesic, anti-inflammatory, or antibiotic medications within the last twelve hours.

Teeth with broken instruments in the canal. Individuals with bruxism problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of different working length measurement methods in endodontic treatment and postoperative pain. | 7 days
  For the purpose of evaluating postoperative pain, the difference between two different working length measurement methods used during endodontic retreatment was analyzed. Postoperative pain was measured by visual analog scale (VAS) scores of the patients during the first 7 days after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)